CLINICAL TRIAL: NCT05301361
Title: Sensitivity of the NIH Toolbox Cognition Battery to Stimulant Treatment in Intellectual Disabilities
Brief Title: Sensitivity of the NIH Toolbox to Stimulant Treatment in Intellectual Disabilities
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 1970634; 5R01HD076189-08 (NIH)
Record Dates: First submitted 2022-03-08; First posted 2022-03-29 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Intellectual Disability; Fragile X Syndrome; Down Syndrome; Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Intellectual Disability; Fragile X Syndrome; Down Syndrome; Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Methylphenidate (Active Comparator)
  Interventions: Drug: Methylphenidate Oral Solution
- Placebo (Placebo Comparator)
  Interventions: Drug: Methylphenidate Oral Solution

INTERVENTIONS:
Drug: Methylphenidate Oral Solution — The XRMPH or matching placebo will be started at a dose of 0.3 mg/kg/day and individually titrated over two weeks. Phone calls at the end of weeks 1, 2, and 3 will be used to collect adverse event and response data. If there is no evidence of side effects and ongoing symptoms of ADHD, the dose will be increased to 0.5 mg/kg/day at one week and 0.7 mg/kg/day at 2 weeks (maximum dose of 60 mg per day consistent with FDA labeled use in youth).

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, crossover trial of extended-release liquid methylphenidate (XRMPH) to evaluate the sensitivity of the NIH Toolbox Cognition Battery (NIHTB-CB) to changes in cognition in children and adolescents ages 6 to 17 with intellectual disability (D) and comorbid Attention Deficit Hyperactivity Disorder (ADHD). The sample will include 68 males or females (expected male: female ratio of 1.8:1 with ID and ADHD as determined by structured diagnostic interview and Conners 3 scores. Additional inclusion criteria will include Full Scale IQ above 50 and mental age greater than or equal to 3 years. In addition, participants must be able to complete NIHTB-CB testing and provide valid scores at baseline. After baseline testing, participants will then be randomized to drug or placebo in a 1:1 ratio (N=34 per group) at the end of the baseline visit. XRMPH in oral suspension supplied as Quillivant XR in 5 mg/ml (Tris Pharma, Monmouth Junction, NJ) will be the active treatment. The XRMPH or matching placebo will be started at a dose of 0.3 mg/kg/day and individually titrated over two weeks. Phone calls at the end of weeks 1, 2, and 3 will be used to collect adverse event and response data. If there is no evidence of side effects and ongoing symptoms of ADHD, the dose will be increased to 0.5 mg/kg/day at one week and 0.7 mg/kg/day at 2 weeks (maximum dose of 60 mg per day consistent with FDA labeled use in youth). The Clinical Global Impression (CGI) will be used as a guide to define optimal dose. If side effects occur the dose will be reduced to the dose level at which there were no side effects. Final optimal dose will be established by the end of week 3 and this will be maintained for 2 weeks until 5 weeks post randomization, at which time the follow-up parent and teacher Conners scales, NIHTB-CB, Go/No-Go, and PedsQL will be completed. Participants will have a washout period of 1 week, will then complete re-assessment at the second baseline, and then will cross over to the other treatment (Quillivant to placebo; placebo to Quillivant), also in a double-blind fashion. In the second treatment arm, patients will have the same titration, monitoring and treatment periods as in the first arm, again followed by repeated assessments at the conclusion of 5 weeks. The accrual of participants and number of visits is shown in the Timeline per 6-month period.

ELIGIBILITY:
Inclusion Criteria:

* IQ below 80
* Mental age 3.0 or higher (Stanford Binet)
* Diagnosis of Intellectual Disability
* Diagnosis of ADHD
* Ability to complete valid NIHTB-CB tests at screening/baseline

Exclusion Criteria:

* stimulant use within 2 weeks prior to randomization
* history of a sensitivity reaction to stimulants
* presence of significant comorbid psychiatric or medical disorder/illness deemed by the site physician as inappropriate for stimulant use (uncontrolled epilepsy, bipolar disorder, psychosis, severe OCD, hypertension, tachycardia hypertension, failure to thrive, psychosis for example)
* a household resident with a current substance abuse disorder

Ages: 6 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-09-29 (Estimated); Study Completion 2026-09-29 (Estimated)

PRIMARY OUTCOMES:
Composite score of NIHTB-CB Flanker, Dimensional Change Card Sort, List Sorting and Speeded Matching tests. | 11 weeks
  The composite score is calculated as the average of the non-age adjusted standard scores of each of these four tests. These standard scores have a mean of 100 and SD of 15. A minimum of 3/4 valid scores is required to calculate an average composite score.

SECONDARY OUTCOMES:
Conners 3 ADHD Rating Scale Inattention Scale | 11 weeks
Conners 3 ADHD Rating Scale Hyperactivity/Impulsivity Scale | 11 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - UC Davis MIND Institute, Sacramento, California
  - Rush University, Chicago, Illinois
  - Cincinnati Children's Hospital, Cincinnati, Ohio